CLINICAL TRIAL: NCT03088046
Title: Circulating Androgen Levels Are Not Affected by the Administration of Vaginal Micronized Progesterone for Withdrawal Bleeding in Patients With Polycystic Ovarian Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Dexeus (Other)
Responsible Party: Principal Investigator, Carlos Dosouto Capel, Fellow in Reproductive Endocrinology, Fundacion Dexeus
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SMD-2017-02
Record Dates: First submitted 2017-03-01; First posted 2017-03-23 (Actual); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Anovulation; Polycystic Ovary Syndrome; Hyperandrogenism
MeSH Terms: conditions — Anovulation; Polycystic Ovary Syndrome; Hyperandrogenism | interventions — Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Micronized Progesterone (Other): Administration of 200 mg of vaginal Micronized Progesterone (100 mg every 12 hours) for a 7-day course
  Interventions: Drug: Micronized Progesterone

INTERVENTIONS:
Drug: Micronized Progesterone — Anovulatory women with Polycystic ovary syndrome and clinical hyperandrogenism attended in our Hospital will participate in the study. A patient information sheet will be provided and written consent will be obtained. Patients who give written consent will participate in the trial. All patient information will be confidential and only be available to researches involved in the study.
  Blood samples will be collected at baseline (Sample #1) and between the 3rd and the 5th day of withdrawal after 7 days of 100mg vaginal MP every 12 hours of administration(Sample#2).

SUMMARY:
Hormonal evaluation of women who are suspected of having Polycystic ovary syndrome (PCOS) involves the measurement of basal levels of androgens and 17-hydroxyprogesterone (17-OHP), which are generally used to establish the presence of hyperandrogenemia. In general, these levels are obtained during the follicular phase to maintain sampling uniformity and avoid spurious increases due to corpus luteum function. However, because most hyperandrogenic patients are oligo/amenorrheic, it is frequently necessary to administer a progestogen to induce withdrawal bleeding and properly time the blood sampling.

Several medications have been described to properly induce withdrawal bleeding , with medroxyprogesterone acetate (MPA) being the most widely use. However, synthetic compounds as MPA do not replicate precisely the constellation of biologic activities of the parent hormone and results in a temporary, albeit clinically relevant, suppression in ovarian function and circulating androgen levels , in addition of several adverse side effects .

In this study, it is hypothesized that the administration of natural progesterone vaginally, which will avoid hepatic first pass, may result in significantly less hormonal suppression.

The authors test this hypothesis by prospectively determining the effect of vaginal micronized progesterone (OMP), administered for the induction of withdrawal bleeding, on the circulating androgen and 17-OHP levels in women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* Chronic ovulatory dysfunction, defined as intermenstrual intervals of >45 days or a total of <8 menstrual cycles per year
* Polycystic ovaries, defined as at least one ovary with >12 follicles between 2 and 9 mm or an ovarian volume >10 mL
* Clinical hyperandrogenism, defined by a Ferriman Gallwey score >8

Exclusion Criteria:

* non-classic congenital adrenal hyperplasia,
* hyperprolactinemia
* thyroid dysfunction
* Oral contraceptives pills taken at least 3 months before the study

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 15 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Change in Total testosterone (TT) | Blood samples will be collected at baseline (Sample #1) , and between the 3rd ad the 5th day of withdrawal after the treatment (sample #2)
  Difference between first and second sample in Total testosterone
Change in free testosterone (FT) | Blood samples will be collected at baseline (Sample #1) , and between the 3rd ad the 5th day of withdrawal after the treatment (sample #2)
  Difference between first and second sample in free testosterone
Change in sex hormone binding globulin (SHBG) | Blood samples will be collected at baseline (Sample #1) , and between the 3rd ad the 5th day of withdrawal after the treatment (sample #2)
  Difference between first and second sample in sex hormone binding globulin (SHBG)
Change in dehydroepiandrosterone sulfate (DHEAS) | Blood samples will be collected at baseline (Sample #1) , and between the 3rd ad the 5th day of withdrawal after the treatment (sample #2)
  Difference between first and second sample in dehydroepiandrosterone sulfate (DHEAS)
Change in androstenedione (A4) | BBlood samples will be collected at baseline (Sample #1) , and between the 3rd ad the 5th day of withdrawal after the treatment (sample #2)
  Difference between first and second sample in androstenedione (A4)
Change in 17-OH progesterone | Blood samples will be collected at baseline (Sample #1) , and between the 3rd ad the 5th day of withdrawal after the treatment (sample #2)
  Difference between first and second sample in 17-OH progesterone

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Livadas S, Boutzios G, Economou F, Alexandraki K, Xyrafis X, Christou M, Zerva A, Karachalios A, Tantalaki E, Diamanti-Kandarakis E. The effect of oral micronized progesterone on hormonal and metabolic parameters in anovulatory patients with polycystic ovary syndrome. Fertil Steril. 2010 Jun;94(1):242-6. doi: 10.1016/j.fertnstert.2009.02.073. Epub 2009 May 5. PMID 19409554
- See also: Related Info — http://www.dexeus.com